CLINICAL TRIAL: NCT03336476
Title: Can Videolaryngoscopy be the First Choice for Tracheal Intubation in Patients With Diabetes
Brief Title: Videolaryngoscopy vs Direct Laryngoscopy for Intubation in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Associate Proffesor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dilek Unal Yazicioglu
Record Dates: First submitted 2017-11-05; First posted 2017-11-08 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus
Keywords: Direct laryngoscopy; Videolaryngoscopy; Diabetes Mellitus; Intubation; Anesthesia
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Prospective randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscopy (Experimental): Videolaryngoscopy the trachea will be intubated using a videolaringoscope
  Interventions: Device: Videolaryngoscopy
- Direct laryngoscopy (Active Comparator): Direct laringoscopy the trachea will be intubated using a laringoscope
  Interventions: Device: Direct laryngoscopy

INTERVENTIONS:
Device: Videolaryngoscopy — Patients will be intubated with the video laryngoscope
  Arms: Videolaryngoscopy
Device: Direct laryngoscopy — Patients will be intubated with the direct laryngoscope
  Arms: Direct laryngoscopy

SUMMARY:
The use of videolarygoscopy (VL) as first choice for tracheal intubation versus direct laryngoscopy (DL) is a matter of debate. These two methods were compared in several studies. Videolaryngoscopes may reduce the number of failed intubations, particularly among patients presenting with a difficult airway. They improve the glottic view and may reduce airway trauma. DM is accepted as a risk factor for difficult intubation. The aim of this study is to compare VL to DL in adult patients requiring tracheal intubation for anesthesia, in terms of intubation success, glottic view quality, intubation failure, intubation time, conversion to another laringoscopy method and adverse outcomes related to tracheal intubation.

DETAILED DESCRIPTION:
The use of videolarygoscopy (VL) as first choice for tracheal intubation versus direct laryngoscopy (DL) is a matter of debate. These two methods were compared in several studies. First attempt intubation success and glottic visualization with VL versus DL by pediatric emergency medicine providers in simulated patients were evaluated and it was concluded that VL was associated with greater first-attempt success during intubation by pediatric emergency physicians on an adult simulator. The ease of viewing the glottis under direct vision during conventional laryngoscopy with the quality of indirectly viewing on a monitor during laryngoscopy with a Macintosh videolaryngoscope was compared in a multicenter study. The results were that VL can lead to better viewing conditions but in rare cases it may result in worse viewing conditions. The study evaluating the efficacy and safety of VL compared to DL in decreasing the time and attempts required and increasing the success rate for endotracheal intubation in neonates concluded that there was insufficient evidence to recommend or refute the use of VL for endotracheal intubation in neonates. Diverse videolaryngoscopes where also compared in patients undergoing tracheal intubation for elective surgery: the GlideScope Ranger (GlideScope, Bothell, WA), the V-MAC Storz Berci DCI (Karl Storz, Tuttlingen, Germany), and the McGrath (McGrath series 5, Aircraft medical, Edinburgh, UK) and tested whether it is feasible to intubate the trachea of patients with indirect videolaryngoscopy without using a stylet. The authors concluded that the trachea of a large proportion of patients with normal airways can be intubated successfully with certain VL blades without using a stylet, although the three studied VL's clearly differ in outcome. The Storz VL displaces soft tissues in the fashion of a classic Macintosh scope, affording room for tracheal tube insertion and limiting the need for stylet use compared with the other two scopes. Although VL's offer several advantages, including better visualization of the glottic entrance and intubation conditions, a good laryngeal view does not guarantee easy or successful tracheal tube insertion. Three different videolarygoscope devices were compared to direct laringoscopy in obese patients undergoing bariatric surgery: Video Mac and GlideScope required fewer intubation attempts that DL and Video Mac provide shorter intubation times and improved glottis view compared to DL. A recent metanalysis stated that videolaryngoscopes may reduce the number of failed intubations, particularly among patients presenting with a difficult airway. They improve the glottic view and may reduce laryngeal/airway trauma. However currently, no evidence indicates that use of a VLS reduces the number of intubation attempts or the incidence of hypoxia or respiratory complications, and no evidence indicates that use of a VL's affects time required for intubation. DM is accepted as a risk factor for difficult intubation.

The aim of this study is to compare VL to DL in adult diabetic patients requiring tracheal intubation for anesthesia, in terms of intubation time, intubation success, glottic view quality, intubation failure, conversion to another laringoscopy method and adverse outcomes related to tracheal intubation.

METHODS After obtaining ethical approval and written informed patient consent, consecutive patients having diabetes mellitus (DM) and requiring elective intubation for anesthesia will be randomly allocated to either the videolaryngoscopy (Group VL) or the direct larngoscopy (Macintosh laryngoscope) (Group DL). Age, gender, body mass index, American Society of Anesthesiologists (ASA) physiologic classification, the duration of DM will be recorded. The patients will be evaluated for difficult airway predictors and the following parameters will be recorded: Malampati class, thyromental distance, sternomental distance, mandibulohyoid distance, interincisor distance, neck circumference, the ability of upper lip overbite and lower lip overbite, the presence of limited neck extension. Fentanyl-propofol-rocuronium will be used for anesthesia induction. After subsequent positive-pressure ventilation using a face mask and an oxygen-air-sevoflurane mixture for 3 min, the trachea will be intubated according to group allocation using either DL (Macintosh laryngoscope) or VL (CMAC). During intubation, the following data will be documented: intubation time, number of intubation attempts, use of extra tools to facilitate intubation, conversion to another laryngoscopy method,intubation difficulty and the quality of the view of the glottis will be assessed according to the Cormack and Lehane scoring system and the percentage of glottic opening. Adverse events related to tracheal intubation will be also evaluated: desaturation (SPO2<94), hypercabia (ETCO2>35), hypertension (mean arterial pressure >20% above baseline values), tachycardia (heart rate >20% above baseline values), new onset arrhythmia, laryngospasm, bronchospasm, airway trauma and sore throat in PACU). The primary outcome measure is the time to intubation; first-attempt intubation success and ease of intubation, secondary outcome measures are the glottic view guality, conversion to another laryngoscopy method and adverse outcomes related to tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery
* Patients needing endotracheal intubation
* Patients having diabetes mellitus

Exclusion Criteria:

* Emergency surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
intubation time | 0-120 seconds after intubation
  The time elapsed between the passage of the larygoscope through the teeth and the detection of ETCO2
first-attempt intubation success rate | first second after intubation
  successful intubation with the allocated device
intubation difficulty | 0-120 seconds after intubation
  number of attempts, number of operators, number of alternative techniques, CL grade, lifting force, laryngeal pressure, position of the vocal cords,

SECONDARY OUTCOMES:
glottic view quality | during laringoscopy
  Cormack Lehane
percentage of glottic opening | during laringoscopy
  the percentage of glottic opening seen, defined by the linear span from the anterior commisure to the interarytenoid notch
the rate of conversion to another laryngoscopy method | 5 seconds after the first attempt to intubate
  the intubation device will be changed if the anesthetist fails to intubate with the allocated device
adverse outcomes related to tracheal intubation. | 1 minute after intubation
  Hypertension, tachycardia, desaturation, hypercarbia, airway trauma, laryngospasm, bronchospasm, sore throat,

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yazicioglu, Assoc Prof, Principal Investigator — Netherlands: Ministry of Health, Welfare and Sports
Locations (1):
- University of Health Sciences Diskapi Yildirim Beyazit Training and Research Hospita, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lingappan K, Arnold JL, Shaw TL, Fernandes CJ, Pammi M. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in neonates. Cochrane Database Syst Rev. 2015 Feb 18;(2):CD009975. doi: 10.1002/14651858.CD009975.pub2. PMID 25691129
- [Result] Donoghue AJ, Ades AM, Nishisaki A, Deutsch ES. Videolaryngoscopy versus direct laryngoscopy in simulated pediatric intubation. Ann Emerg Med. 2013 Mar;61(3):271-7. doi: 10.1016/j.annemergmed.2012.09.008. Epub 2012 Oct 18. PMID 23083969
- [Result] van Zundert A, Maassen R, Lee R, Willems R, Timmerman M, Siemonsma M, Buise M, Wiepking M. A Macintosh laryngoscope blade for videolaryngoscopy reduces stylet use in patients with normal airways. Anesth Analg. 2009 Sep;109(3):825-31. doi: 10.1213/ane.0b013e3181ae39db. PMID 19690253
- [Result] Hofstetter C, Scheller B, Flondor M, Gerig HJ, Heidegger T, Brambrink A, Thierbach A, Wilhelm W, Wrobel M, Zwissler B. [Videolaryngoscopy versus direct laryngoscopy for elective endotracheal intubation]. Anaesthesist. 2006 May;55(5):535-40. doi: 10.1007/s00101-006-0998-3. German. PMID 16688385
- [Result] Lewis SR, Butler AR, Parker J, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation. Cochrane Database Syst Rev. 2016 Nov 15;11(11):CD011136. doi: 10.1002/14651858.CD011136.pub2. PMID 27844477